CLINICAL TRIAL: NCT02972411
Title: Controlled Hyperventilation as Prophylaxis for Acute Mountain Sickness: A Randomized Controlled Trial
Brief Title: Controlled Hyperventilation as Prophylaxis for Acute Mountain Sickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Trabajador de Santiago (Other)
Responsible Party: Principal Investigator, Sebastián Drago Pérez, Orthopaedic Surgeon, Hospital del Trabajador de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HospitalTS
Record Dates: First submitted 2016-10-25; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Altitude Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Voluntary increase in respiration
  Interventions: Behavioral: Voluntary ventilatory response
- Acetazolamide (Active Comparator): Administration of Acetazolamide 125mg. since 24 hours before ascent and until 48 hours post altitude exposure, and absence of altitude sickness symptoms
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Behavioral: Voluntary ventilatory response — Training of the subjects for voluntary increase in the respiratory minute ventilation
  Arms: Intervention
Drug: Acetazolamide — Acetazolamide 125mg. PO every 12 hours since 24 hours before ascent, until 48 hours at high altitude
  Arms: Acetazolamide

SUMMARY:
This study evaluates the safety and efficacy of the voluntary ventilatory response as prophylaxis for acute mountain sickness, measured by the Lake Louise Self-Report Score, comparing to a group using acetazolamide.

DETAILED DESCRIPTION:
Rationale: Acute mountain sickness (AMS) is a common condition among people who go to altitude and stay at altitude. Acclimatization is the most important mechanism in order to reduce the risk of AMS, however, this is not possible or adequate in a large part of the cases. Recently, there are indications that adjustment of respiration by means of a voluntary increase in the respiratory minute volume can have a similar prophylactic effect. The purpose of this study is to measure the effect of the voluntary increase of the minute volume by means of controlled hyperventilation as prophylaxis for acute mountain sickness without prior acclimatization, with AMS being expressed in the Lake Louise Self-Report Score (LLSRS).

Objective: To investigate the safety and efficacy of the voluntary increase in minute ventilation by means of controlled hyperventilation as prophylaxis for AMS, measured by the LLSRS in a randomized controlled trial ascending to 4954m altitude.

Study design: Prospective randomized controlled trial, safety and efficacy.

Study population: 30 healthy subjects

Intervention: The investigational prophylaxis is controlled hyperventilation. Participants in the interventional group will be trained to hyperventilate in a controlled fashion doing a series of exercises during the 4 days prior to the ascent. They will also be taught in a practical way to recognize early clinical signs and symptoms of hypocapnia.

Main study parameters/endpoints: Safety and efficacy measured by comparing the LLSRS between the two groups. Target end-tidal CO2 ( PETCO2) will be measured to objectify adequate hyperventilation. Symptoms of hypocapnia due to the (pre-)intervention as well as any adverse events will be reported and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Living at lower altitude than 900 meters

Exclusion Criteria:

* Cardiac or pulmonary comorbidity
* Smoking
* Infectious disease during the last 30 days
* BMI> 30
* Pharmaceutical use as diuretics, corticosteroids, acetazolamide, or anti -inflammatory drugs during the 2 weeks prior to the study
* A history of high altitude cerebral edema or high altitude pulmonary edema
* Cardiovascular risk factors such as a personal history of cardiovascular disease, familial history of major adverse cardiovascular events (MACE) at age younger than 45 yrs, hypercholesterolemia and stroke.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Lake Louise Score | Up to 5 months
  Intensity and prevalence of Acute Mountain Sickness. During Ascent.

SECONDARY OUTCOMES:
PETCO2 | Up to 5 months
  Pressure of expired CO2, measured with a monitor in the moutain. During ascent.
Pulse oxygen saturation | Up to 5 months
  During ascent.
Respiratory rate | Up to 5 months
  During ascent
Heart rate | Up to 5 months
  During ascent
Borg Scale | Up to 5 months
  During ascent

OTHER OUTCOMES:
Training satisfactory. PETCO2 below 20 mmHg | Up to 6 months
  After ascent.
Training satisfactory after Ascent. PETCO2 below 20mmHg | Up to 6 months
  After ascent.
hypoxic ventilatory response | Up to 6 months
  Before ascent

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Drago, MD, Principal Investigator — Hospital del Trabajador Santiago
Locations (1):
- 110 Sports and health center, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartsch P, Swenson ER. Clinical practice: Acute high-altitude illnesses. N Engl J Med. 2013 Jun 13;368(24):2294-302. doi: 10.1056/NEJMcp1214870. PMID 23758234
- [Background] Buijze GA, Hopman MT. Controlled hyperventilation after training may accelerate altitude acclimatization. Wilderness Environ Med. 2014 Dec;25(4):484-6. doi: 10.1016/j.wem.2014.04.009. Epub 2014 Oct 14. No abstract available. PMID 25443751
- [Background] Luks AM, McIntosh SE, Grissom CK, Auerbach PS, Rodway GW, Schoene RB, Zafren K, Hackett PH; Wilderness Medical Society. Wilderness Medical Society consensus guidelines for the prevention and treatment of acute altitude illness. Wilderness Environ Med. 2010 Jun;21(2):146-55. doi: 10.1016/j.wem.2010.03.002. Epub 2010 Mar 10. PMID 20591379
- [Background] Richalet JP, Larmignat P, Poitrine E, Letournel M, Canoui-Poitrine F. Physiological risk factors for severe high-altitude illness: a prospective cohort study. Am J Respir Crit Care Med. 2012 Jan 15;185(2):192-8. doi: 10.1164/rccm.201108-1396OC. Epub 2011 Oct 27. PMID 22071330
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Vargas M, Osorio J, Jimenez D, Moraga F, Sepulveda M, Del Solar J, Hudson C, Cortes G, Leon A. [Acute mountain sickness at 3500 and 4250 m. A study of symptom, incidence and severity]. Rev Med Chil. 2001 Feb;129(2):166-72. Spanish. PMID 11351468
- [Background] Acetazolamide in control of acute mountain sickness. Lancet. 1981 Jan 24;1(8213):180-3. PMID 6109857
- [Background] Bernardi L, Passino C, Spadacini G, Bonfichi M, Arcaini L, Malcovati L, Bandinelli G, Schneider A, Keyl C, Feil P, Greene RE, Bernasconi C. Reduced hypoxic ventilatory response with preserved blood oxygenation in yoga trainees and Himalayan Buddhist monks at altitude: evidence of a different adaptive strategy? Eur J Appl Physiol. 2007 Mar;99(5):511-8. doi: 10.1007/s00421-006-0373-8. Epub 2007 Jan 6. PMID 17206440
- [Background] Bernardi L, Schneider A, Pomidori L, Paolucci E, Cogo A. Hypoxic ventilatory response in successful extreme altitude climbers. Eur Respir J. 2006 Jan;27(1):165-71. doi: 10.1183/09031936.06.00015805. PMID 16387950
- [Background] Moore LG, Harrison GL, McCullough RE, McCullough RG, Micco AJ, Tucker A, Weil JV, Reeves JT. Low acute hypoxic ventilatory response and hypoxic depression in acute altitude sickness. J Appl Physiol (1985). 1986 Apr;60(4):1407-12. doi: 10.1152/jappl.1986.60.4.1407. PMID 3084449